CLINICAL TRIAL: NCT04850144
Title: Comparison of Tiotropium Pharmacokinetics After Inhalation From Tiotropium Easyhaler® Product Variants and After Spiriva® Capsules Administered Via HandiHaler®; Study in Healthy Volunteers
Brief Title: Pharmacokinetic Study Comparing Tiotropium Easyhaler® and Spiriva® HandiHaler®
Acronym: TESSA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 3122005
Record Dates: First submitted 2021-04-13; First posted 2021-04-20 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Charcoal

STUDY DESIGN:
Intervention Model Description: The study is a 2-part 4-period crossover study where the study subjects participate either in part 1 (20 subjects) or in part 2 (20 subjects). Parts can run in sequence or parallel. All study subjects receive single dose of Tiotropium Easyhaler on 3 periods and Spiriva HandiHaler on 1 period.
Masking Description: Bioanalytical laboratory will be blinded with regard to the sequence of the product administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Tiotropium Easyhaler Product variant D (Experimental)
  Interventions: Drug: Tiotropium Bromide Monohydrate
- Tiotropium Easyhaler Product variant E (Experimental)
  Interventions: Drug: Tiotropium Bromide Monohydrate
- Tiotropium Easyhaler Product variant F (Experimental)
  Interventions: Drug: Tiotropium Bromide Monohydrate
- Tiotropium Easyhaler Product variant G (Experimental)
  Interventions: Drug: Tiotropium Bromide Monohydrate
- Tiotropium Easyhaler Product variant H (Experimental)
  Interventions: Drug: Tiotropium Bromide Monohydrate
- Spiriva HandiHaler (Active Comparator)
  Interventions: Drug: Tiotropium Bromide Monohydrate
- Tiotropium Easyhaler Product variant F administered with oral activated charcoal (Experimental)
  Interventions: Drug: Tiotropium Bromide Monohydrate; Drug: Tiotropium Easyhaler with oral activated charcoal

INTERVENTIONS:
Drug: Tiotropium Bromide Monohydrate — Tiotropium Easyhaler 10 µg/dose Product variant D
  Arms: Tiotropium Easyhaler Product variant D
Drug: Tiotropium Bromide Monohydrate — Tiotropium Easyhaler 10 µg/dose Product variant E
  Arms: Tiotropium Easyhaler Product variant E
Drug: Tiotropium Bromide Monohydrate — Tiotropium Easyhaler 10 µg/dose Product variant F
  Arms: Tiotropium Easyhaler Product variant F; Tiotropium Easyhaler Product variant F administered with oral activated charcoal
Drug: Tiotropium Bromide Monohydrate — Tiotropium Easyhaler 10 µg/dose Product variant G
  Arms: Tiotropium Easyhaler Product variant G
Drug: Tiotropium Bromide Monohydrate — Tiotropium Easyhaler 10 µg/dose Product variant H
  Arms: Tiotropium Easyhaler Product variant H
Drug: Tiotropium Bromide Monohydrate — Spiriva 18 µg/capsule inhaled via Handihaler
  Arms: Spiriva HandiHaler
Drug: Tiotropium Easyhaler with oral activated charcoal — The charcoal suspension will be administered orally with Tiotropium Easyhaler 10 µg/dose Product variant F
  Arms: Tiotropium Easyhaler Product variant F administered with oral activated charcoal

SUMMARY:
Absorption of inhaled tiotropium is compared between five Tiotropium Easyhaler product variants and Spiriva capsules inhaled via HandiHaler without charcoal. Absorption of tiotropium is compared between one Easyhaler product variant administered with and without charcoal.

ELIGIBILITY:
Main inclusion criteria:

1. Healthy males and females
2. 18-60 years of age
3. Body mass index 19-30 kg/m2
4. Weight at least 50 kg
5. Written informed consent obtained

Main exclusion criteria:

1. Evidence of a clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic, endocrine, neurological or psychiatric disease
2. Any condition requiring regular concomitant treatment
3. Any clinically significant abnormal laboratory value or physical finding that in the opinion of the investigator could interfere with the interpretation of study results or cause a health risk for the subject
4. Known hypersensitivity to tiotropium bromide, atropine or its derivatives or lactose
5. Pregnant or lactating females and females of childbearing potential not using contraception of acceptable effectiveness
6. Blood donation or loss of significant amount of blood within 90 days prior to the first study treatment administration.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Peak tiotropium concentration in plasma (Cmax) | between 0-72 hours after dosing
Area under the concentration-time curve from time zero to 30 minutes (AUC30 minutes) | 0-30 minutes after dosing
Area under the concentration-time curve from time zero to 72 hours (AUC72 hours) | 0-72 hours after dosing

SECONDARY OUTCOMES:
Time to reach peak concentration in plasma (tmax) | between 0-72 hours after dosing

OTHER OUTCOMES:
Adverse events | througout the study, an average 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Orion Corporation Clinical Study Director, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- Clinical Pharmacology Unit, Orion Corporation, Espoo, Finland

IPD SHARING:
Plan to Share IPD: No